CLINICAL TRIAL: NCT06043011
Title: Clinical Research Platform on Treatment, Quality of Life and Outcome of Patients With Hematologic Malignancies (RUBIN) - Extension of Tumor Registry Lymphatic Neoplasms
Brief Title: Registry Platform Hematologic Malignancies (RUBIN) - Extension of Tumor Registry Lymphatic Neoplasms
Acronym: RUBIN
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-080485
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Diffuse Large B-cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL); Waldenström's Macroglobulinemia (WM)
Keywords: non-Hodgkin lymphoma (NHL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Chronic Lymphocytic Leukemia (CLL): Patients with CLL receiving systemic treatment (physician's choice)
  Interventions: Other: Routine care as per site standard.
- Diffuse Large B-cell Lymphoma (DLBCL): Patients with DLBCL receiving systemic treatment (physician's choice)
  Interventions: Other: Routine care as per site standard.
- Follicular Lymphoma (FL): Patients with FL receiving systemic treatment (physician's choice)
  Interventions: Other: Routine care as per site standard.
- Mantle Cell Lymphoma (MCL): Patients with MCL receiving systemic treatment (physician's choice)
  Interventions: Other: Routine care as per site standard.
- Marginal Zone Lymphoma (MZL): Patients with MZL receiving systemic treatment (physician's choice)
  Interventions: Other: Routine care as per site standard.
- Waldenström's macroglobulinemia (WM): Patients with WM receiving systemic treatment (physician's choice)
  Interventions: Other: Routine care as per site standard.

INTERVENTIONS:
Other: Routine care as per site standard. — Physician's choice according to patient's needs.

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter registry platform to document uniform data on characteristics, molecular diagnostics, treatment and course of disease, to collect patient-reported outcomes and to establish a decentralized biobank for patients with hematological malignancies in Germany.

DETAILED DESCRIPTION:
RUBIN is a national, observational, prospective, longitudinal, multicenter registry platform with the purpose to record information on the antineoplastic treatment of hematological malignancies in Germany.

It will identify common therapeutic sequences and changes in the treatment of the disease, and will analyse the impact of novel treatments on the outcome of patients in routine care. Unmet needs and areas with the potential for improvement in routine care are to be identified.

At inclusion, data in patient characteristics, comorbidities, clinical characteristics and previous treatments, if applicable, are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and clinical outcome are documented.

Health-realted quality of life in patients with hematological malignancies will be evaluated for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of the respective NHL
* If patient is alive: signed written informed consent

  * For patients participating in the PRO survey: IC prior to or at day of start of respective line of treatment.
  * For patients not participating in the PRO survey: IC latest eight weeks after start of respective line of treatment.

Exclusion Criteria:

* No systemic therapy for respective lymphoid malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with hematologic malignancies requiring systemic treatment
Sampling Method: Probability Sample
Enrollment: 2950 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality) | 5 years
  Documentation of anamnestic data and therapy sequences. Documentation of anamnestic data and therapy sequences

SECONDARY OUTCOMES:
Best Response | 5 years
  Documentation of response rates per line of treatment.
Progression-free survival | 5 years
  Documentation of progression-free survival per line of treatment.
Overall survival | 5 years
  Documentation of overall survival time.
Health-related quality of life (Patient-reported outcome) | 1 year
  EORTC QLQ-C30 core questionnaire
Disease-specific quality of life (Patient-reported outcome, patients with CLL) | 1 year
  EORTC QLQ-CLL17
Disease-specific quality of life (Patient-reported outcome, patients with LG-NHL) | 1 year
  EORTC QLQ-NHL-LG20
Disease-specific quality of life (Patient-reported outcome, patients with HG-NHL) | 1 year
  EORTC QLQ-NHL-HG29

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Claus, Prof. Dr., Study Chair — Universitätsklinikum Augsburg, Germany; Tobias Dechow, Study Chair — Studienzentrum Onkologie Ravensburg, Germany; Paul Graf La Rosée, Prof. Dr., Study Chair — Schwarzwald-Baar Klinikum, Germany; Jens Kisro, Dr., Study Chair — Lübecker Onkologische Schwerpunktpraxis, Germany; Patrick Marschner, Dr., Study Chair — Praxis für Interdisziplinäre Hämatologie und Onkologie, Freiburg, Germany; Ingo Tamm, PD Dr., Study Chair — Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin, Germany; Robert Zeiser, Prof. Dr., Study Chair — Universitätsklinikum Freiburg, Germany
Locations (1):
- Praxis für Interdisziplinäre Hämatologie und Onkologie, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No